CLINICAL TRIAL: NCT02643888
Title: Identification of Pre-existing Kinase Domain Mutations in Subclones of Ph-positive Leukemias
Brief Title: Pre-existing Kinase Domain Mutations in Ph-positive Leukemias
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Anna Kinderkrebsforschung (Other)
Collaborators: Medical University of Vienna (Other); National Research Center for Radiation Medicine in Kiev (Unknown); St. Petersburg State Pavlov Medical University (Other); UHKT Prague (Unknown)
Responsible Party: Principal Investigator, Prof DDr Thomas Lion, Medical Director, St. Anna Kinderkrebsforschung
Other Study IDs: BCR-ABL 001
Record Dates: First submitted 2015-10-30; First posted 2015-12-31 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA samples from CML patients obtained from bone marrow/peripheral blood and fingernail clippings
Oversight: Data Monitoring Committee: No

SUMMARY:
The main task of this study includes analyses of the BCR-ABL1 (breakpoint cluster region/Abelson) gene and mutations in the BCR-ABL1 tyrosine kinase domain within flow-sorted stem cells from the bone marrow and/or peripheral blood specimens. To assess the germline configuration of the patient, DNA from fingernail clippings will be investigated.

DETAILED DESCRIPTION:
Background Single or multiple point mutations in the tyrosine kinase domain (TKD) of the BCR-ABL1 fusion gene in chronic myeloid leukemia (CML) and Ph-chromosome positive acute lymphoblastic leukemia represent the most important known mechanism of resistance to tyrosine kinase inhibitors (TKIs). It is conceivable that pre-existing point mutations in CML stem cells attributable to the genomic instability conferred by the BCR-ABL1 fusion protein give rise to the outgrowth of resistant subclones and onset of treatment-insensitive disease under the selection pressure of TKI therapy. Early detection of such subclones may therefore be of prognostic and therapeutic relevance. The recently published immunophenotype of CML stem cells (Hermann et al. Blood 2014), and our recent report on an NGS (next-generation sequencing)-based method facilitating sensitive detection and quantitative monitoring of BCR-ABL1 subclones carrying single or compound mutations (Kastner et al. European Journal of Cancer 2014) facilitate the screening for clinically relevant mutant subclones in stem cells or early progenitor cells.

Hypothesis Detection of mutant subclones within the stem cell or early progenitor compartments at diagnosis or early into therapy of Ph-positive leukemias, and monitoring of their proliferation kinetics, permit early prediction of resistant disease under the ongoing TKI treatment.

Experimental approach Bone marrow (BM) and peripheral blood (PB) samples will be collected upon informed consent from patients with Ph-positive leukemia at diagnosis (BM+PB), and subsequently at 3-month intervals (PB;BM upon availability) during the first year of therapy based on or including TKIs. Isolation of CD (cluster of differentiation) 34+ cells carrying additional phenotypic markers characterizing stem cells or early progenitor cells (CD38-/CD25+/CD26+ in CML, CD19 in Ph-ALL) will be performed by flow sorting. The entire BCR-ABL1 tyrosine kinase domain (TKD) will be amplified from cDNA (complementary DNA) or specific exons of interest from DNA by established protocols, and bidirectional sequencing will be performed by ultra-deep sequencing using NGS. Mutant subclones identified at diagnosis or after debulking of most of the treatment-sensitive leukemic burden early into treatment (3 month time point), will be monitored by NGS until month 12 of therapy. BCR-ABL1 transcripts will be monitored according to the International Scale (IS) in parallel. DNA isolated from fingernail clippings will be used as germline control for the ABL1 TKD. The testing will be performed in a blinded fashion to prevent treatment adjustments according to experimental data.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Ph-positive leukemia

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study plan includes 30 adult patients with Ph-positive leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2023-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Leukemic stem/progenitor cells defined by a specific marker profile will be isolated from BM/PB by flow sorting. Screening for and monitoring of BCR-ABL1 TKD mutant subclones at the cDNA/DNA levels within the 1st year of TKI therapy will be done by NGS. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lion, MD PhD Prof, Principal Investigator — Children´s Cancer Research Institute
Locations (1):
- Medical Universitiy of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Preuner S, Danzer M, Proll J, Potschger U, Lawitschka A, Gabriel C, Lion T. High-quality DNA from fingernails for genetic analysis. J Mol Diagn. 2014 Jul;16(4):459-66. doi: 10.1016/j.jmoldx.2014.02.004. Epub 2014 Apr 30. PMID 24795088
- [Background] Preuner S, Mitterbauer G, Mannhalter C, Herndlhofer S, Sperr WR, Valent P, Lion T. Quantitative monitoring of BCR/ABL1 mutants for surveillance of subclone-evolution, -expansion, and -depletion in chronic myeloid leukaemia. Eur J Cancer. 2012 Jan;48(2):233-6. doi: 10.1016/j.ejca.2011.08.015. Epub 2011 Sep 28. PMID 21955823
- [Background] Preuner S, Denk D, Frommlet F, Nesslboeck M, Lion T. Quantitative monitoring of cell clones carrying point mutations in the BCR-ABL tyrosine kinase domain by ligation-dependent polymerase chain reaction (LD-PCR). Leukemia. 2008 Oct;22(10):1956-61. doi: 10.1038/leu.2008.97. Epub 2008 Apr 24. No abstract available. PMID 18432261